CLINICAL TRIAL: NCT00876551
Title: Endoscopic - Vacuum Assisted Closure of Intrathoracic Postsurgical Leaks
Brief Title: Endoscopic-vacuum Assisted Closure of Intrathoracic Postsurgical Leaks
Acronym: EVACoIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Dr. Jochen Wedemeyer, Department of Gastroenterology, Hepatology and Endocrinology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Spongebop01
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2009-04

CONDITIONS: Mediastinitis; Esophageal Neoplasms; Anastomotic Leakage
Keywords: Negative-Pressure Wound Therapy; Endoscopic/endoluminal V.A.C. therapy; Esophagectomy; Anastomotic leakage; Anastomosis, Surgical
MeSH Terms: conditions — Mediastinitis; Esophageal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- E-V.A.C. (Experimental): Patients that are treated with E-V.A.C.
  Interventions: Procedure: Endoscopic vacuum assisted closure

INTERVENTIONS:
Procedure: Endoscopic vacuum assisted closure — 1. Endoscopic debridement of wound using a regular biopsy forceps.
  2. Introduction via the nose and oral exteriorization of a silicone duodenal tube (Freka Tube, 15 Ch, Fresenius Kabi, Bad Homburg v.d. H. Germany)
  3. Fixation of a polyurethane foam (sponge, pore size 400-600 µm, KCI, Wiesbaden Germany) to the tip of the duodenal tube with a mersilene suture (0,35mm, Johnson & Johnson, St-Stevens-Woluwe, Belgium).
  4. Trimming of the sponge to the specific wound size.
  5. Endoscopic placement of the sponge in the intrathoracic leak with a grasping forceps (Olympus, Germany)
  6. Application of continuous suction of 125mmHg using vacuum pump (KCI, Wiesbaden Germany).
  7. Sponge exchange twice a week until wound grounds are clean and closed
  Other Names: Endoluminal vacuum assisted closure; E-V.A.C.; Endosponnge

SUMMARY:
The purpose of this study is to determine the short and long term outcome of endoscopic vacuum assisted closure of intrathoracic postsurgical leaks.

DETAILED DESCRIPTION:
Intrathoracic leakage is a serious complication after esophageal surgery. The reported incidence of esophageal anastomotic leaks after gastrectomy and esophagectomy ranges from 5% to almost 30%. Within the last 10 years endoscopic treatment has changed the approach to intrathoracic anastomotic leakages. Application of metal clips, injection of fibrin glue and placement of self expanding metal or plastic stents (SEMS/SEPS) have been reported to successfully achieve closure of postoperative anastomotic leaks in approximately 66-100%. Alternative endoscopically treatment modalities are welcome especially in cases of failure of the above mentioned endoscopic treatment modalities to prevent the necessity of surgical reintervention which is associated with high mortality or mutilating surgical outcome such as proximal diversion with cervical esophagostomy.

Vacuum-assisted closure (V.A.C.) is an established treatment modality for extensive cutaneous infected wounds. The V.A.C. system device is based on a negative pressure applied to the wound via a vacuum sealed sponge tissue. The sponge results in formation of granulation tissue, while the vacuum removes wound secretions and reduces edema and therefore improves blood flow, all together achieving consecutive wound closure. Since its introduction in the late 1990´s the number of indications for the V.A.C. system has steadily increased. Recently the endoluminal application of a vacuum assisted wound closure system for the closure of rectal anastomotic fistulas has been reported. Our group reported the successful closure of intrathoracic anastomotic leaks in two cases by endoscopic placement of a vacuum assisted closure system. Here we plan to study the efficacy, safety and long term outcome of E-V.A.C. to treat major intrathoracic postsurgical leaks.

ELIGIBILITY:
Inclusion Criteria:

* All patients at the Medical School Hannover that present with intrathoracic postsurgical leakage that can be intubated with a regular 9.2mm diameter endoscope (Olympus GIF-165, Olympus
* Age over 18 years old
* Signed informed consent

Exclusion Criteria:

* Small leakage that can be treated with clips
* Refusal to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Closure of postsurgical leak | 6 weeks

SECONDARY OUTCOMES:
Short term complications | 6 weeks
Long term complications | 6 months
number of endoscopic interventions | 6 weeks
time to leak closure | 6 weeks
C reactive protein | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Wedemeyer, MD, Principal Investigator — Dept. of Gastroenterology, Hepatology and Endocrinology, Medical School Hannover
Locations (1):
- Dept. of Gastroenterology, Hepatology and Endocrinology, Medical School Hannover, Hanover, Germany

REFERENCES:
- [Background] Wedemeyer J, Schneider A, Manns MP, Jackobs S. Endoscopic vacuum-assisted closure of upper intestinal anastomotic leaks. Gastrointest Endosc. 2008 Apr;67(4):708-11. doi: 10.1016/j.gie.2007.10.064. PMID 18374029
- [Derived] Wedemeyer J, Brangewitz M, Kubicka S, Jackobs S, Winkler M, Neipp M, Klempnauer J, Manns MP, Schneider AS. Management of major postsurgical gastroesophageal intrathoracic leaks with an endoscopic vacuum-assisted closure system. Gastrointest Endosc. 2010 Feb;71(2):382-6. doi: 10.1016/j.gie.2009.07.011. Epub 2009 Oct 30. PMID 19879566